CLINICAL TRIAL: NCT00245765
Title: Multicenter, Dose Response, Randomized, Double Blind, Parallel, Placebo Controlled Clinical Trial to Evaluate the Efficacy and the Safety of Subcutaneous CDP870 in Subjects Suffering From Moderate-to-severe Chronic Plaque Psoriasis Who Are Candidates for Systemic Therapy and/or Phototherapy and/or Photochemotherapy
Brief Title: Efficacy Study of CDP870 in Subjects With Chronic Plaque Psoriasis Who Are Candidate for Systemic Therapy and/or Phototherapy/Photochemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C87040; 2005-002141-39 (EudraCT Number)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: chronic plaque psoriasis, anti TNFα; CDP870, Cimzia
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Subcutaneous injections of Placebo every 2 weeks
  Interventions: Other: Placebo
- Certolizumab Pegol 200 mg (Experimental): Subcutaneous injections of 400 mg initial dose at week 0 with 200 mg every 2 weeks thereafter
  Interventions: Drug: Certolizumab Pegol
- Certolizumab Pegol 400 mg (Experimental): Subcutaneous injections of 400 mg every 2 weeks
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — * Pharmaceutical Form: solution for injection in pre-filled syringe
  * Route of Administration: subcutaneous use
  Other Names: Cimzia
  Arms: Certolizumab Pegol 200 mg; Certolizumab Pegol 400 mg
Other: Placebo — Matching Placebo to Certolizumab Pegol
  Arms: Placebo

SUMMARY:
A study to assess the safety and efficacy of 2 different doses of CDP870 versus placebo, administered during 12 weeks, to patients suffering from moderate to severe chronic plaque psoriasis, extended by a 12 to 24 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women > 18 years
* Subjects with chronic plaque psoriasis stable for at least 3 months and moderate to severe for at least 6 months
* Subjects with Psoriasis Area and Severity Index (PASI) ≥ 12 and Body Surface Area (BSA) ≥ 10 %
* Subjects were candidates for systemic psoriasis therapy and/or phototherapy and/or photochemotherapy

Exclusion Criteria:

* Subjects with an erythrodermic, guttate, palmar or plantar, generalized pustular form of psoriasis
* A history of chronic infection, recent serious or life-threatening infection (within six months, including herpes zoster), or any current sign or symptom that may indicate an infection (e.g. fever, cough);
* White blood cell counts less than 4000/mm^3 or more than 20000/mm^3
* Suspected or diagnosed demyelinating disease of the central nervous system (e.g. multiple sclerosis or optic neuritis)
* Systemic Lupus
* Non respect of adequate wash out periods for treatments that might have an impact on the disease
* Any associated disease that could be impacted by the study treatment intake
* Any other condition, which in the Investigator's judgment would make the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (15):
- France (6):
  - Besançon
  - Créteil
  - Nice
  - Paris
  - Pierre-Bénite
  - Saint-Etienne
- Germany (9):
  - Berlin
  - Bonn
  - Essen
  - Frankfurt
  - Göttingen
  - Hamburg
  - Kiel
  - Mainz
  - Münster

REFERENCES:
- [Result] Ortonne JP, Tasset C, Reich K. Efficacy of certolizumab pegol, a PEGylated Fab' fragment of an anti-alpha monoclonal antibody, in patients previously exposed to biologicals: preliminary results of a randomised, placebo-controlled, phase II clinical trial in psoriasis. J.Eur.Acad.Dermatol.Venereol. 22[Suppl 1], 2007. Vienna, 16th Congress of the European Academy of Dermatology and Venereology (EADV), May 16-20, 2007.
- [Result] Ortonne JP, Sterry W, Tasset C, Reich K. Safety and efficacy of subcutaneous certolizumab pegol, a new anti-TNF-alpha monoclonal antibody, in patients with moderate-to-severe chronic plaque psoriasis: preliminary results from a double-blind, placebo-controlled trial. J.Am.Acad.Dermatol. 56[Suppl 2], AB6. 2007. Washington, DC, 65th Annual Meeting of the American Academy of Dermatology (AAAD), February 2-7, 2007.
- [Result] Reich K, Tasset C, Ortonne J. Efficacy and safety of certolizumab pegol, in patients with chronic plaque psoriasis: preliminary results of a randomized, double-blind, placebo-controlled trial. Ann.Rheum.Dis. 66[Suppl 2], 251. 2007. Barcelona, Annual European Congress of Rheumatology EULAR 2007, June 13-16, 2007.
- [Result] Ortonne JP, Sterry W, Tasset C, Reich K. Certolizumab pegol, the first pegylated anti-TNF alpha, is effective and well tolerated in patients with moderate-to-severe chronic plaque psoriasis: preliminary data from a phase II study. J.Eur.Acad.Dermatol.Venereol. 21[Suppl 1], 26. 2007. Rhodes, Greece, 15th Congress of the European Academy of Dermatology and Venereology (EADV), October 4-8, 2006.
- [Result] Ortonne JP, Sterry W, Coteur G, Keininger DL, Reich K. Improved health-related quality of life in psoriasis patients following 10 weeks' treatment with certolizumab pegol: data from a Phase II study. 2007. Buenos Aires, Argentina, 21st World Congress of Dermatology, October 1-5, 2007.
- [Result] Reich K, Sterry W, Tasset C, Terpstra I, Ortonne JP. Efficacy and time to relapse with certolizumab pegol, the first pegylated anti-TNF alpha agent, in patients with moderate-to-severe chronic plaque psoriasis: Phase II study results. 2007. Buenos Aires, Argentina, 21st World Congress of Dermatology, October 1-5, 2007.
- [Result] Ortonne JP, Reich K, Sterry W, Terpstra I. Safety and efficacy (PASI 90 and global evaluation) of subcutaneous certolizumab pegol in patients with moderate to severe chronic plaque psoriasis: Results from a double-blind, placebo-controlled trial. J.Am.Acad.Dermatol. 58[Suppl 2], AB4. 2008. San Antonio, 66th Annual Meeting of the American Academy of Dermatology (AAD), February 1-5, 2008.
- [Result] Ortonne JP, Reich K, Keininger DL. Certolizumab pegol improved health-related quality of life in patients with psoriasis: Data from a phase II study. J.Am.Acad.Dermatol. 58[Suppl 2], AB121. 2008. San Antonio, 66th Annual Meeting of the American Academy of Dermatology (AAD), February 1-5, 2008.
- [Result] Reich K, Ortonne JP, Gottlieb AB, Terpstra IJ, Coteur G, Tasset C, Mease P. Successful treatment of moderate to severe plaque psoriasis with the PEGylated Fab' certolizumab pegol: results of a phase II randomized, placebo-controlled trial with a re-treatment extension. Br J Dermatol. 2012 Jul;167(1):180-90. doi: 10.1111/j.1365-2133.2012.10941.x. Epub 2012 Jun 11. PMID 22413944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in October 2005 and concluded in November 2006.
Pre-assignment Details: The study included a 12-week Treatment Period and a 12 to 24-week Follow-up Period. Participant Flow refers to the Intention-to-treat Set.
Groups:
- Placebo (ITT): Subcutaneous injections of Placebo every 2 weeks
- Certolizumab Pegol 200 mg (ITT): Subcutaneous injections of 400 mg initial dose at week 0 with 200 mg every 2 weeks thereafter
- Certolizumab Pegol 400 mg (ITT): Subcutaneous injections of 400 mg every 2 weeks
Period: Overall Study
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Started | 59 | 59 | 58
Safety Population (The safety population consisted of all subjects who were exposed to study medication.) | 58 (One subject in the Placebo (PBO) group received one injection of CDP870 200 mg on one occasion.) | 60 (For safety analysis, the PBO group subj. who received CDP870 was considered to be in the 200mg group) | 57 (One subject in the 400 mg group was randomized by mistake but did not receive study medication.)
Completed | 27 | 45 | 50
Not Completed | 32 | 14 | 8
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 14 | 7 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Other reason | 2 | 0 | 1
Not completed — Other | 13 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-To-Treat (ITT) population consisting of all randomized subjects.
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT) | Total Title
Number analyzed (Participants) | 59 | 59 | 58 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 57 | 55 | 166
  >=65 years | 5 | 2 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.30 (12.78) | 43.26 (10.12) | 43.64 (12.36) | 43.40 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 16 | 53
  Male | 37 | 44 | 42 | 123

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Psoriasis Activity and Severity Index (PASI75) Response at Week 12
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI75 response at Week 12 is defined as a decrease in PASI score at Week 12 from Baseline of at least 75 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
percentage of subjects | 6.8 | 74.6 | 82.8
Statistical Analysis 1: Comparison: Placebo (ITT) vs Certolizumab Pegol 200 mg (ITT); Test type: Superiority; p < 0.001, Regression, Logistic; Logistic regression with treatment and baseline severity of psoriasis as factors; Odds Ratio (OR) = 40.2, 95% CI 2-sided [13.7 to 150.3] — Confidence limits are based on likelihood ratio statistics
Statistical Analysis 2: Comparison: Placebo (ITT) vs Certolizumab Pegol 400 mg (ITT); Test type: Superiority; p < 0.001, Regression, Logistic; Logistic regression with treatment and baseline severity of psoriasis as factors; Odds Ratio (OR) = 73.4, 95% CI 2-sided [23.5 to 292.6] — Confidence limits are based on likelihood ratio statistics

2. Primary Outcome: Achievement of a Physician's Global Assessment (PGA) of Clear or Almost Clear at Week 12
Description: The overall severity of the disease was evaluated using the following 6-point scale:
  5 = Severe: Very marked plaque elevation, scaling, and/or erythema. 4 = Moderate to severe: Marked plaque elevation, scaling, and/or erythema. 3 = Moderate: Moderate plaque elevation, scaling, and/or erythema. 2 = Mild: Slight plaque elevation, scaling, and/or erythema
  1 = Almost clear: Intermediate between mild and clear 0 = Clear: No signs of psoriasis (post-inflammatory hyperpigmentation may be present)
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
percentage of subjects | 1.7 | 52.5 | 72.4
Statistical Analysis 1: Comparison: Placebo (ITT) vs Certolizumab Pegol 200 mg (ITT); Test type: Superiority; p < 0.001, Regression, Logistic; Logistic regression with treatment and baseline severity of psoriasis as factors. Confidence limits are based on likelihood ratio statistics; Odds Ratio (OR) = 64.1, 95% CI 2-sided [12.7 to 1169.1]
Statistical Analysis 2: Comparison: Placebo (ITT) vs Certolizumab Pegol 400 mg (ITT); Test type: Superiority; p < 0.001, Regression, Logistic; Logistic regression with treatment and baseline severity of psoriasis as factors; Odds Ratio (OR) = 162.6, 95% CI 2-sided [31.4 to 2999.2] — Confidence limits are based on likelihood ratio statistics

3. Secondary Outcome: Time to Psoriasis Activity and Severity Index 50 (PASI50)
Description: Time to PASI50 is defined as the time elapsed between the start of the Treatment Period (Week 0) and the first occurrence of PASI50 during the Treatment Period.
  This variable is defined only for those patients who have achieved PASI75 at the end of the Treatment Period (Week 12).
Time Frame: During the 12-weeks Treatment Period
Population: Only those subjects from the Intention-To-Treat (ITT) population who are PASI75 responder at Week 12 are included in the analysis of this variable.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 4 | 44 | 48
days | 56.50 [14.00 to 99.00] | 21.00 [20.00 to 28.00] | 22.00 [21.00 to 30.00]

4. Secondary Outcome: Time to Psoriasis Activity and Severity Index 75 (PASI75)
Description: Time to PASI75 is defined as the time elapsed between the start of the Treatment Period (Week 0) and the first occurrence of PASI75 during the Treatment Period.
  This variable is defined only for those patients who have achieved PASI75 at the end of the Treatment Period (Week 12).
Time Frame: During the 12-weeks Treatment Period
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 4 | 44 | 48
days | 77.50 [42.00 to 99.00] | 42.50 [28.00 to 56.00] | 55.50 [42.00 to 69.00]

5. Secondary Outcome: Time to Relapse
Description: Time to relapse is defined as the time elapsed between the last dose and when maximal improvement in PASI from Baseline was reduced by > 50 %. This variable is defined only for those patients who have achieved PASI75 at the end of the Treatment Period (Week 12).
Time Frame: During the 12-weeks Treatment Period
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 4 | 44 | 48
weeks | NA [NA to NA] — This parameter applied only to those subjects who had achieved PASI75 at the end of the treatment period and who had an event of relapse. | 22.14 [17.00 to 26.00] | 20.14 [17.00 to 22.29]

6. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI50) Response at Week 12
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI50 response at Week 12 is defined as a decrease in PASI score at Week 12 from Baseline of at least 50 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
percentage of subjects | 11.9 | 86.4 | 93.1

7. Secondary Outcome: Achievement of a Psoriasis Activity and Severity Index (PASI90) Response at Week 12
Description: Determining the PASI score involves the evaluation of erythema, infiltration, and desquamation and body surface area involvement over 4 body regions. These regions are the head, trunk, upper and lower extremities.
  PASI90 response at Week 12 is defined as a decrease in PASI score at Week 12 from Baseline of at least 90 %.
Time Frame: Week 12
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
percentage of subjects | 1.7 | 39.0 | 46.6

8. Secondary Outcome: Experience of a Rebound Effect Within 2 Months After Stopping Therapy
Description: Rebound is defined as worsening of psoriasis over baseline value with more than 125 % or new pustular, erythrodermic or more inflammatory psoriasis within 2 months of stopping therapy.
Time Frame: Within 2 months of stopping therapy
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
percentage of subjects | 15.3 | 1.7 | 1.7

9. Secondary Outcome: Percent of Body Surface Area (BSA) Affected by Psoriasis at Week 12
Description: Two methods were used for the evaluation of BSA:
  1. The area of one side of a subject's flat closed hand was used to represent 1 % to the total body surface area (BSA) to estimate the extent of skin involvement in subjects with psoriasis
  2. The rule of nines method assumed that the total BSA comprises head (9 %), anterior trunk (upper, 9 %; lower, 9 %), posterior trunk (upper, 9 %; lower, 9 %), each leg (anterior, 9 %; posterior, 9 %), each arm (9 %) and genitalia (1 %)
Time Frame: Week 12
Population: ITT population consisting of all randomized subjects. The analysis was performed for week 12 using observed case data (i.e., no imputation was performed for missing data). By week 12, there were 29 patients who had prematurely discontinued the study.
Measure: Mean (Standard Deviation); unit: percentage of affected Body Surface Area
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 40 | 53 | 54
percentage of affected Body Surface Area | 28.8 (17.2) | 7.1 (9.3) | 5.6 (6.5)

10. Secondary Outcome: Absolute Change From Baseline in the Body Surface Area (BSA) Affected by Psoriasis at Week 12
Description: Two methods were used for the evaluation of BSA:
  1. The area of one side of a subject's flat closed hand was used to represent 1 % to the total body surface area (BSA) to estimate the extent of skin involvement in subjects with psoriasis
  2. The rule of nines method assumed that the total BSA comprises head (9 %), anterior trunk (upper, 9 %; lower, 9 %), posterior trunk (upper, 9 %; lower, 9 %), each leg (anterior, 9 %; posterior, 9 %), each arm (9 %) and genitalia (1 %) A positive value in Change from Baseline indicates an improvement from Baseline. The higher the positive value, the higher the change.
Time Frame: Baseline up to Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percent of total Body surface area
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 40 | 53 | 54
Percent of total Body surface area | 3.2 (11.9) | 18.3 (15.1) | 22.6 (15.7)

11. Secondary Outcome: Time to Discontinuation From the Treatment Period Due to Lack of Efficacy or Worsening of Psoriasis
Time Frame: During the 12-week Treatment Period
Population: Intention-To-Treat (ITT) population consisting of all randomized subjects.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo (ITT) | Certolizumab Pegol 200 mg (ITT) | Certolizumab Pegol 400 mg (ITT)
Number analyzed (Participants) | 59 | 59 | 58
days | 42.0 [21.0 to 75.0] | 59.5 [35.0 to 70.0] | 49.0 [21.0 to 77.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline (Week 0) over the 12-weeks Treatment Period until the end of the Follow-up Period (up to 36 weeks).
Description: The safety population consisted of all subjects who were exposed to study medication. One subject in the PBO group received one injection of CDP870 200 mg on one occasion. In the safety analysis, this subject was considered to be in the 200 mg group. One subject in the 400 mg group was randomized by mistake but did not receive study medication. This subject discontinued from the study due to an adverse event. This subject was randomized and is part of the ITT population.
Groups:
- Placebo (SS): Subcutaneous injections of Placebo every 2 weeks
- Certolizumab Pegol 200 mg (SS): Subcutaneous injections of 400 mg initial dose at week 0 with 200 mg every 2 weeks thereafter
- Certolizumab Pegol 400 mg (SS): Subcutaneous injections of 400 mg every 2 weeks
Arm/Group | Placebo (SS) | Certolizumab Pegol 200 mg (SS) | Certolizumab Pegol 400 mg (SS)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/58 | 2/60 | 5/57
Other Adverse Events (participants affected / at risk) | 34/58 | 32/60 | 27/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SS) (N=58) | Certolizumab Pegol 200 mg (SS) (N=60) | Certolizumab Pegol 400 mg (SS) (N=57)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (SS) (N=58) | Certolizumab Pegol 200 mg (SS) (N=60) | Certolizumab Pegol 400 mg (SS) (N=57)
Constipation (Gastrointestinal disorders) | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 1
Asthenia (General disorders) | 3 | 3 | 3
Chills (General disorders) | 3 | 1 | 1
Fatigue (General disorders) | 0 | 4 | 0
Injection site haematoma (General disorders) | 0 | 4 | 2
Injection site irritation (General disorders) | 0 | 3 | 1
Pyrexia (General disorders) | 3 | 2 | 4
Bronchitis (Infections and infestations) | 3 | 0 | 4
Herpes simplex (Infections and infestations) | 1 | 4 | 0
Influenza (Infections and infestations) | 4 | 2 | 2
Nasopharyngitis (Infections and infestations) | 10 | 4 | 12
Rhinitis (Infections and infestations) | 4 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 2
Headache (Nervous system disorders) | 9 | 13 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days